CLINICAL TRIAL: NCT06936202
Title: Effects of Spirulina Supplementation on Mental Health in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Senior Associate Dean, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00021993
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Depression; Mental Acuity
Keywords: spirulina; depression; mental acuity
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This is a parallel arm, 8-week, randomized controlled study with an experimental arm and a control arm.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spirulina capsules (Experimental): six capsules daily (totaling 3 g)
  Interventions: Other: Spirulina capsules
- Placebo (Placebo Comparator): Pea powder - 6 capsules daily
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Spirulina capsules — active intervention
  Arms: spirulina capsules
Other: Placebo — no active ingredient
  Arms: Placebo

SUMMARY:
Spirulina platensis is a form of cyanobacteria, a blue-green algae, and is a superfood most known for being rich in protein, vitamins and minerals, and healthful phytochemicals. Spirulina supports brain health through neuroprotection offered by its antioxidants, anti-inflammatory properties, and hormone regulation.

The aim of this study is to supplement healthy adults from a campus community with 3g of spirulina, daily, for 8 weeks to improve mood and mental acuity in comparison to receiving a placebo.

DETAILED DESCRIPTION:
Spirulina is nutrient-dense with vitamins and minerals which provide antioxidants and anti-inflammatory mechanisms to help reduce oxidative stress and ROS activity. Preclinical studies have indicated Spirulina can reduce inflammatory cytokines, such as IL-1β, and reverse stress responses and oxidative damage in BDNF, nuclear factor erythroid 2-related factor (NRF2), and ultimately the phosphorylation of protein-kinase B (AKT), which promotes cell growth. In addition to these benefits, fatty acids, gamma-linolenic acid (GLA) and glycolipids, support gut health and the immune system. In combination, all these nutrients help increase neuroprotection and brain health.

It is evident that Spirulina supports brain health through neuroprotection, antioxidants, anti-inflammatory properties, and hormone regulation. Research supports Spirulina reversing neurodegenerative diseases due to several of these beneficial properties. There have been many studies that utilize Spirulina to improve cognitive function in Alzheimer's Disease, Parkinson's Disease, ulcerative colitis, IBD, fibromyalgia and even in TBI and Ischemic stroke.

Although many of these diseases have depressive symptoms, few of these studies have evaluated the impact of Spirulina on mood. Furthermore, no studies have been conducted relating depression and the cyanobacteria. It is possible that Spirulina supplements can be used to reduce feelings of hopelessness and lack of energy, by providing additional vitamins, minerals, amino acids, and fatty acids, on a daily basis. This study aims to compare spirulina and its improvement on mood, in health college students, by daily supplementation of 3g of Spirulina over a span of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* ages 18-65
* no underlying chronic disease or acute conditions
* no autoimmune conditions
* do not consume alcohol in excess, smoke, use recreational drugs
* does not follow restrictive diets
* will be recruited from the ASU university campus.

Exclusion Criteria:

* not have been clinically diagnosed with depression
* not taking antidepressants, anxiety, or stress medications, or any other medications
* drugs, or supplements that could influence mental capacities
* not pregnant or breastfeeding
* not a competitive athlete

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
POMS (profile of mood states questionnaire) | conducted at baseline and at week 8 (study's end)
  A validated measure consisting of 65 brief phrases, asking how they have personally felt over the last week, including today. The participants were asked to carefully rate their response on a 5-point Likert scale, ranging from 'not at all' to 'extremely'.
Trail Making Test | conducted at baseline and at week 8 (study's end)
  The TMT consists of two iterations - versions A and B - and brief samples of each will be provided for the participant to practice prior to the longer, scored version. This is a timed paper and pencil test requiring the participant to connect a series of numbers and/or letters that are randomly arranged.

CONTACTS AND LOCATIONS:
Locations (1):
- 850 PBC, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to publish in ICMJE journals